CLINICAL TRIAL: NCT06303505
Title: A First-in-human Dose Escalation and Optimization Phase I/IIa Study to Investigate Safety, Tolerability, PK, and Efficacy of the NaPi2b ADC TUB-040 in Patients With Platinum-resistant High-grade Ovarian Cancer (PROC) or r/r Adenocarcinoma Non-small Cell Lung Cancer (NSCLC)
Brief Title: FiH Study to Investigate Safety, PK and Efficacy of the NaPi2b ADC TUB-040 in Patients With PROC or r/r Adenocarcinoma NSCLC
Acronym: NAPISTAR1-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tubulis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NAPISTAR 1-01; 2024-511074-80 (EudraCT Number)
Record Dates: First submitted 2024-02-06; First posted 2024-03-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Non-small Cell Lung Cancer
Keywords: TUB-040; ADC; PROC
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Platinum resistant ovarian cancer (Experimental)
  Interventions: Drug: TUB-040
- Non small cell lung cancer-adenocarcinoma (Experimental)
  Interventions: Drug: TUB-040

INTERVENTIONS:
Drug: TUB-040 — A complete treatment cycle is defined as 21 calendar days. TUB-040 will be administered as an intravenous (IV) solution on day 1 of each treatment cycle

SUMMARY:
The purpose of this multicentric, open label trial (NAPISTAR 1-01) is to evaluate the safety/tolerability, pharmacokinetics and preliminary efficacy of TUB-040 and to find the best dose of TUB-040 in patients with ovarian cancer and Non Small Cell Lung Cancer. TUB-040 is an antibody-drug-conjugate which delivers a topoisomerase I inhibitor to tumor cells which overexpress the target NaPi2b. The study consists of two parts: In dose escalation, ovarian cancer patients and lung cancer patients receive increasing doses of TUB-040 until the maximal tolerated dose is found. In dose optimization, at least two doses are compared with each other to determine which dose is optimal for patients.

TUB-040 is given IV every 3 weeks until the disease progresses or the patient has to stop due to side effects.

ELIGIBILITY:
Inclusion Criteria (for all patients)

1. Male or non-pregnant, non-breastfeeding female, age 18 years or older at the date of consent.
2. Disease not amenable to curative intent treatment.
3. Patients have exhausted the standard of care treatment (SoC) with expected survival benefit and are not denied SoC with expected survival benefit by participating in the trial.
4. Radiologically measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, that includes at least 1 lesion not previously irradiated.
5. Eastern Cooperative Oncology Group (ECOG) 0-1.
6. Have a life expectancy of more than 12 weeks for disease-related mortality, as evaluated by the INV.
7. Patients must be willing to sign an archival tissue release form for research purposes and determination of biomarker (eg NaPi2b) expression.
8. Patients must be willing to undergo a non-contrast high resolution computed tomography (HRCT) of the thorax scan and pulmonary function testing (PFT) at screening.
9. Adequate organ function
10. Resolution of all acute toxic effects of prior therapy or surgical procedures to ≤grade 1 (except alopecia, hyperpigmentation, or discoloration (incl. vitiligo) of the skin and nails, stable immune-related toxicity such as hypothyroidism on hormone replacement, adrenal insufficiency on ≤10 mg daily prednisone [or equivalent], chronic grade 2 peripheral sensory neuropathy after prior taxane therapy).
11. Patients of childbearing potential (FCBP) who are sexually active with a non-sterilized partner must use at least one highly effective method of contraception from the time of screening and must agree to continue using such precautions until the end of exposure, plus 5 half-lives and 6 months add-on in the case of patients assigned female at birth. Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the patient for the duration of the study treatment and the above-referred period after the end of the exposure. Periodic abstinence (e.g., calendar ovulation, symptothermal, post-ovulation methods), the rhythm method, and the withdrawal method are not acceptable methods of contraception.
12. In the opinion of the investigator, the patient must be able to understand, give written informed consent, and comply with all study-related procedures, medication use, and evaluations.
13. The patient must not have a history of non-compliance with medical regimens or be considered potentially unreliable and/or uncooperative.
14. The patient must be willing to sign and date the informed consent form (ICF)

Exclusion Criteria (for all patients)

1. The patient is pregnant, lactating or breastfeeding or has a positive serum pregnancy test during the screening period.
2. History of hypersensitivity to exatecan or excipients of the TUB-040 formulation, including ADCs with deruxtecan, exatecan or camptothecan as a payload.
3. Disease that is refractory to topoisomerase-I inhibitors, defined as progression during or within 6 months of the last infusion.
4. Patients are not allowed to participate in interventional clinical studies either concurrently or within the previous 28 days or within 5 half-lives of any investigational pharmacologic agents or imaging materials, including dyes, investigational surgical techniques, or devices.
5. Patients with spinal cord compression or active central nervous system disease.
6. Prior radiotherapy <2 weeks from trial inclusion.
7. Major surgery within 21 days prior to signing the ICF, unless the patient is recovered at that time.
8. Has a history of non-infectious ILD/pneumonitis/radiation pneumonitis that required steroids or has current ILD/pneumonitis.
9. Has an oxygen saturation of <93% on room air at rest.
10. Has a forced vital capacity of <60% and diffusing capacity of the lung for carbon monoxide <70%.
11. Has a QTcF >470 ms
12. History of nephrotic syndrome
13. Active corneal disease, or history of corneal disease within 12 months prior to enrollment.
14. Active, uncontrolled impairment of the urogenital, renal, hepatobiliary, cardiovascular, gastrointestinal, neurologic, or hematopoietic systems which, in the opinion of the investigator, would predispose the patient to the development of complications from the administration of protocol therapy.
15. History of another malignancy with ongoing treatment or not yet free from disease for 2 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or other malignancy with a similar expected curative outcome.
16. Documented other concurrent non-malignant comorbidities such as unstable or uncontrolled pectoral angina, myocardial infarction during the last 6 months, valvular heart disease that requires treatment, acute myocarditis, or congestive heart failure (CHF) (New York Heart Association III or IV).
17. Any concurrent chemotherapy, radiotherapy (except for local radiation therapy of lesions that may cause imminent complications), immunotherapy, or corticoid therapy.
18. Live vaccines within 30 days prior to study entry.
19. Patients with acute or chronic infections such as:

    1. Patients who are HBsAg positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks and have an undetectable HBV viral load prior to randomization.
    2. Patients with a history of HCV infection are eligible if HCV viral load is undetectable at screening.
    3. HIV infected patients must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease
    4. Any other known unresolved and active bacterial, viral, fungal, mycobacterial, or other infection at screening.
    5. History of severe and recurrent infections per INV judgment.
    6. History of progressive multifocal leukoencephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Determination of MTD | From enrollment until 30 days after last study drug
  The highest dose is defined at which no more than 1 of 3 patients have had a Dose Limiting Toxicity (DLT) according to NCI CTCAE V5.0 criteria

SECONDARY OUTCOMES:
Maximum plasma/serum concentration (Cmax) | From enrollment until 30 days after last study drug
  The concentration of TUB-040 (conjugated ADC), total mAb, and free payload (Cmax will be derived).
Through plasma/serum concentration (Cmin) | From enrollment until 30 days after last study drug
  The concentration of TUB-040 (conjugated ADC), total mAb, and free payload (Cmin will be derived).
The time taken to reach the maximum concentration (Tmax) | From enrollment until 30 days after last study drug
  The concentration of TUB-040 (conjugated ADC), total mAb, and free payload (Tmax will be derived).
Area Under Curve (AUC) | From enrollment until 30 days after last study drug
  The concentration of TUB-040 (conjugated ADC), total mAb, and free payload (AUC will be derived).
Half life (T1/2) | From enrollment until 30 days after last study drug
  The concentration of TUB-040 (conjugated ADC), total mAb, and free payload (T1/2 will be derived).
Determination of immunogenicity | From enrollment until 30 days after last study drug
  Number and percentage of patients developing anti-TUB-040 antibodies, and semiquantitative titer assessment. It is measured at cycles 1, 2, 3, 4, 6, 8, 10, post treatment
Determination of efficacy | From enrollment until 30 days after last study drug
  ORR by investigator assest Recist 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Fingerle-Rowson, MD, PhD, Study Director — Tubulis GmbH
Locations (14):
- United States (6):
  - Mount Sinai, New York, New York
  - Christ Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Next Oncology Dallas, Irving, Texas
  - Next Oncology Virginia, Fairfax, Virginia
- UZ Leuven, Leuven, Belgium
- Germany (2):
  - Charité Universitätsmedizin Berlin, Berlin
  - University Hospital Cologne Department of Internal Medicine I, Cologne
- Arensia Exploratory Medicine, Cluj-Napoca, Romania
- Spain (2):
  - Clínica universidad de Navarra, Madrid
  - NEXT Oncology Madrid, Madrid
- Arensia Exploratory Medicine, Kyiv, Ukraine
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
we first want to evaluate the ICMJE Guidelines